CLINICAL TRIAL: NCT02921763
Title: Duphaston® Tablets 5 mg - A Survey on Efficacy and Safety in Patients With Endometriosis
Brief Title: A Survey on Efficacy and Safety in Patients With Endometriosis
Status: Completed | Type: Observational
Sponsor: Mylan Inc. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: DUPKST16002
Record Dates: First submitted 2016-09-13; First posted 2016-10-03 (Estimated); Results first posted 2022-06-13 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Dydrogesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dydrogesterone: Dydrogesterone 20 mg (4 tablets) per day should be orally administered in 2 divided doses (in the morning and evening). It should be administered for 21 days; dosage starts on the 5th day of each menstrual cycle until 25th day. The administration period will be from the start of Duphaston treatment (cycle 1) to cycle 4.
  Interventions: Drug: Dydrogesterone

INTERVENTIONS:
Drug: Dydrogesterone
  Other Names: Duphaston

SUMMARY:
This survey is intended to collect efficacy and safety data of Duphaston® Tablets in patients with endometriosis under actual condition of its use and to obtain data for effectively and safely utilizing this drug.

DETAILED DESCRIPTION:
In Japan, Duphaston® Tablets have appeared in 1965 for the treatment of endometriosis and been used at some medical institutions. However, after releasing of danazol in the early 1980's and gonadotropin-releasing hormone (GnRH) agonists in the late 1980's, pseudomenopause therapy became mainstream because of its high efficacy. However, pseudopregnancy therapy was recognized again due to adverse reactions associated with pseudomenopause therapy. After 2000, low-dose estrogen/progestin (LEP) combination drugs (as LEP products, ethinylestradiol/norethisterone combination drug and ethinylestradiol/drospirenone combination drug) and dienogest have been utilized as drugs that are safer and can be administered for a long time. In recent years, Duphaston® Tablets are increasing recognized again from the viewpoints of its efficacy and safety because the drug has no effect to inhibit ovulation or effect on basal body temperature, a diagnosis of ovulation and other conditions may be made by following up basal body temperature, and pregnancy may be achieved even during treatment with Duphaston. As previously mentioned, Duphaston® Tablets are an old drug, and there are only few clinical data from Japanese patients; thus, its latest clinical efficacy and safety data are being demanded again mainly by obstetrician-gynecologists.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to < 50 years
* Subjects with a chocolate cyst of the ovary measuring 3 cm in diameter on transvaginal ultrasonography at patient enrollment
* Subjects with a menstrual cycle of 25 to 38 days who ovulate and are confirmed to have normal menstruation at patient enrollment

Exclusion Criteria:

* Subjects who used GnRH agonists within 6 months before patient enrollment
* Subjects who utilized hormone preparations containing corpus luteum hormone or estrogen as an active ingredient, low-dose contraceptive pills, middle-dose contraceptive pills, testosterone derivatives, or herbal products indicated for endometriosis within 3 months before patient enrollment
* Subjects who received surgical treatment for endometriosis such as transvaginal alcohol fixation, laparotomy or laparoscopic surgery within 2 months before patient enrollment
* Subjects who are pregnant or may possibly be pregnant at patient enrollment
* Subjects who are in breast feeding at patient enrollment
* Subjects who are determined by the investigator/subinvestigator to be not suitable for the subjects of the survey because of other reasons
* Subjects with liver disorder or liver disease
* Subjects with known hypersensitivity to the active substance or to any of the excipients
* Subjects with known or suspected progestogen dependent neoplasms (e.g. meningioma)
* Subjects with undiagnosed vaginal bleeding
* Subjects with a past or current history of heart or kidney disease
* Subjects with porphyria
* Subjects with depression
* Subjects with abnormal liver function values caused by acute or chronic liver disease
* Subjects with rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucosegalactose malabsorption

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects of the survey will be patients with a diagnosis of endometriosis.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2017-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jo Kitawaki, MD., PhD., Principal Investigator — Kyoto Prefectural University of Medicine
Locations (15):
- Japan (15):
  - Mylan Investigational Site G, Tokyo, Chiyodaku
  - Mylan Investigational Site N, Tokyo, Chuouku
  - Mylan Investigational Site C, Kyoto, Fushimiku
  - Mylan Investigational Site D, Saitama, Iwatsukiku
  - Mylan Investigational Site M, Okayama, Kurashikishi
  - Mylan Investigational Site H, Kyoto, Kyotanabeshi
  - Mylan Investigational Site A, Kamigyō-ku, Kyoto
  - Mylan Investigational Site I, Kyoto, Nakagyoku
  - Mylan Investigational Site K, Kyoto, Nakagyoku
  - Mylan Investigational Site F, Kyoto, Nakagyoku
  - Mylan Investigational Site J, Tokyo, Shibuyaku
  - Mylan Investigational Site B, Bunkyō, Tokyo
  - Mylan Investigational Site E, Kyoto, Ukyouku
  - Mylan Investigational Site L, Kyoto, Yosanocho
  - Mylan Investigational Site O, Tokushima

IPD SHARING:
Plan to Share IPD: Undecided
We will consider after completion of CSR

REFERENCES:
- [Derived] Kitawaki J, Koga K, Kanzo T, Momoeda M. An assessment of the efficacy and safety of dydrogesterone in women with ovarian endometrioma: An open-label multicenter clinical study. Reprod Med Biol. 2021 Jun 4;20(3):345-351. doi: 10.1002/rmb2.12391. eCollection 2021 Jul. PMID 34262403

RESULTS

PARTICIPANT FLOW:
Groups:
- Dydrogesterone: Dydrogesterone 20 mg (4 tablets) per day should be orally administered in 2 divided doses (in the morning and evening). It should be administered for 21 days; dosage starts on the 5th day of each menstrual cycle until 25th day. The administration period will be from the start of Duphaston treatment (cycle 1) to cycle 4.
  Dydrogesterone
Period: Overall Study
Arm/Group | Dydrogesterone
Started | 60
Completed | 42
Not Completed | 18
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 4
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1
Not completed — No data obtained | 2

BASELINE CHARACTERISTICS:
Population: Of 60 subjects whose case report forms were collected, 59 subjects were included in the "safety analysis set," after excluding one subject (reason: one subject, no data entered).
Arm/Group | Dydrogesterone
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (7.0)
Age, Customized [Count of Participants; unit: Participants]
  >= 20 and < 30 years old | 11
  >= 30 and < 40 years old | 21
  >= 40 and < 50 years old | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 59
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 59
Height [Mean (Standard Deviation); unit: cm] — Population: the corresponding data has not been acquired
  cm
    number analyzed (Participants) | 56
    (all) | 159.8 (5.0)
Weight [Mean (Standard Deviation); unit: kg] — Population: the corresponding data has not been acquired
  kg
    number analyzed (Participants) | 56
    (all) | 54.4 (9.3)
Menstrual cycle [Mean (Standard Deviation); unit: days] | 28.6 (2.3)
History of surgical treatment (for endometriosis) [Count of Participants; unit: Participants]
  No | 48
  Yes | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in the Volume of Ovarian Chocolate Cyst (If There Are Two or More Cysts, a Total Volume)
Description: In measurement of ovarian chocolate cyst, on a section visualizing the maximum diameter, two radial directions, namely the maximum diameter (D1) and maximum diameter (D2) orthogonal to D1, will be measured. A chocolate cyst of the ovary will be deemed as a spheroid, and its volume will be calculated using the following formula: [(D1 + D2) × 1/2]3 × 0.52 (π = 3.1). If there are two or more chocolate cysts of the ovary, similarly, two radial directions (D1 and D2) of each cyst will be measured. Also, each of their volumes will be calculated in the same manner.
  The change rate within ±15% from the total volume measured before treatment was defined as "unchanged," and the rate out of this range was defined as "decreased" or "increased."
Time Frame: Before treatment initiation (baseline), 3 months, and 5 months.
Population: 57 subjects were included in the efficacy analysis set. Of 57 subjects in the efficacy analysis set, changes in the volume of ovarian chocolate cyst before and after treatment in 52 subjects with values before and after Duphaston treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dydrogesterone
Number analyzed (Participants) | 52
Participants
  Decreased | 26
  Unchanged | 13
  Increased | 13
Statistical Analysis 1: Comparison: Dydrogesterone; For the volume calculated from the major and minor axes of ovarian chocolate cyst, the values before treatment initiation and at last observation were compared, frequency of increase and decrease was summarized and the sign test was performed separately in the "efficacy analysis set" and "study completers."; Test type: Superiority; p = 0.0533, Sign test

2. Primary Outcome: Volume of Ovarian Chocolate Cyst Over Time (If There Are Two or More Cysts, a Total Volume)
Description: In measurement of ovarian chocolate cyst, on a section visualizing the maximum diameter, two radial directions, namely the maximum diameter (D1) and maximum diameter (D2) orthogonal to D1, will be measured. A chocolate cyst of the ovary will be deemed as a spheroid, and its volume will be calculated using the following formula: [(D1 + D2) × 1/2]3 × 0.52 (π = 3.1). If there are two or more chocolate cysts of the ovary, similarly, two radial directions (D1 and D2) of each cyst will be measured. Also, each of their volumes will be calculated in the same manner.
Time Frame: Before treatment initiation (baseline), 3 months, and 5 months.
Population: Of the safety analysis set (59 subjects), 57 subjects were included in the "efficacy analysis set," after excluding twe subjects (reason: one subject, use of concomitant medication indicated for endometriosis; one subject, violation of entry criteria).
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Dydrogesterone
Number analyzed (Participants) | 57
cm^3
  Cycle -1 | 45.76 (40.70)
  Cycle 3: number analyzed (Participants) | 39
  Cycle 3 | 51.97 (50.20)
  Cycle 5: number analyzed (Participants) | 40
  Cycle 5 | 60.27 (109.04)

3. Primary Outcome: Volume of Ovarian Chocolate Cyst Over Time (If There Are Two or More Cysts, a Total Volume), Absolute Change From Baseline
Description: The absolute change from baseline were calculated on an individual basis and these were totalled and means ± SD calculated.
  For the mean value of the absolute changes shown here, the mean value of the absolute changes of the cases that could be measured at each time point is calculated. In other words, of the 57 cases with the volume value of baseline, Cycle 3 calculates the mean value of the absolute change in 39 cases with the volume value at this time, and Cycle 5 calculates the mean value of the absolute change in 40 cases with the volume value at this time.
  The remaining 18 cases are excluded from this calculation because there is no volume value for Cycle 3 and the absolute change from baseline cannot be calculated. The same applies to the 17 cases of Cycle 5.
  For this reason, these values cannot be calculated directly from the volume mean value at each time point shown in the result measurement 2.
Time Frame: Before treatment initiation (baseline), 3 months, and 5 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^3
Groups:
- Cycle 3: 2 Cycles of dydrogesterone treatment completed
- Cycle 5: 4 Cycles of dydrogesterone treatment completed (at the completion of the observation period)
Arm/Group | Cycle 3 | Cycle 5
Number analyzed (Participants) | 39 | 40
cm^3 | 0.04 (24.91) | 8.48 (83.69)
Statistical Analysis 1: Comparison: Cycle 3; For the volume calculated from the major and minor axes of ovarian chocolate cyst (a total volume if there were two or more cysts), the value, difference from the value before treatment and change rate were calculated using the summary statistics at each measurement point and last observation in each analysis set, namely "efficacy analysis set" and "study completers," and the Wilcoxon signed-rank test was performed for the difference and change rate; Test type: Superiority; p = 0.7328, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cycle 5; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1193, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Volume of Ovarian Chocolate Cyst Over Time (If There Are Two or More Cysts, a Total Volume), % Change From Baseline
Description: The % change from baseline were calculated on an individual basis and these were totalled and means ± SD calculated.
  For the mean value of the % changes shown here, the mean value of the % changes of the cases that could be measured at each time point is calculated. In other words, of the 57 cases with the volume value of baseline, Cycle 3 calculates the mean value of the % change in 39 cases with the volume value at this time, and Cycle 5 calculates the mean value of the % change in 40 cases with the volume value at this time.
  The remaining 18 cases are excluded from this calculation because there is no volume value for Cycle 3 and the % change from baseline cannot be calculated. The same applies to the 17 cases of Cycle 5.
  For this reason, these values cannot be calculated directly from the volume mean value at each time point shown in the result measurement 2.
Time Frame: Before treatment initiation (baseline), 3 months, and 5 months.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cycle 3 | Cycle 5
Number analyzed (Participants) | 39 | 40
percent change | 3.97 (46.06) | -6.40 (86.88)
Statistical Analysis 1: Comparison: Cycle 3; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.7221, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cycle 5; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0861, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change Over Time in Dysmenorrhea Score (Total of the Dysmenorrhea Severity Score and the Analgesic Use Score)
Description: The dysmenorrhea score is the sum of the dysmenorrhea severity score and the analgesic use score. Shown as the mean value for the number of cases at each time point.
  A dysmenorrhea severity score is defined as follows. None: Score 0, Rarely interfering with work (study and house work): Score 1, Interfering with work (study and house work) requiring lying down to rest: Score 2, Being confined to bed for 1 day, being unable to work (study and house work): Score 3.
  A analgesic use score is defined as follows. None: Score 0, An analgesic was used for a day during the last (or current) menstruation period: Score 1, An analgesic was used for 2 days during the last (or current) menstruation period: Score 2, An analgesic was used for 3 days during the last (or current) menstruation period: Score 3 The minimum dysmenorrhea score is 0 and the maximum dysmenorrhea score is 6.
Time Frame: Baseline, 1 month, 2 months, 3 months, 4 months, and 5 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cycle -1: Before treatment initiation (Baseline)
- Cycle 1: At treatment initiation (the administration could be started during menstruation of cycle 1)
- Cycle 2: 1 Cycles of dydrogesterone treatment completed
- Cycle 4: 3 Cycles of dydrogesterone treatment completed
Arm/Group | Cycle -1 | Cycle 1 | Cycle 2 | Cycle 3 | Cycle 4 | Cycle 5
Number analyzed (Participants) | 57 | 57 | 52 | 50 | 45 | 42
score on a scale | 2.30 (1.89) | 1.75 (1.83) | 1.31 (1.67) | 1.12 (1.42) | 1.00 (1.38) | 1.05 (1.40)

6. Secondary Outcome: Change Over Time in Visual Analogue Scale (VAS) for Dysmenorrhea
Description: A straight line with a total length of 10 cm was prepared. This straight line was defined as "no pain" at the left end and "Worst pain imaginable" at the right end.
  The cases marked the degree of pain on this straight line at each time point, and the length (cm) from the left end of the line (0) was measured.
  The minimum value of VAS is 0 cm (no pain) and the maximum value is 10 cm (Worst pain imaginable).
  The units on a scale is "cm".
Time Frame: Baseline, 1 month, 2 months, 3 months, 4 months, and 5 months.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cycle -1 | Cycle 1 | Cycle 2 | Cycle 3 | Cycle 4 | Cycle 5
Number analyzed (Participants) | 55 | 53 | 41 | 43 | 39 | 35
cm | 4.33 (2.92) | 3.35 (2.66) | 2.54 (2.36) | 2.37 (2.41) | 2.03 (2.39) | 2.01 (2.26)

7. Secondary Outcome: Change in Serum CA125
Description: CA-125 is a glycoprotein antigen recognized by the monoclonal antibody OC125 made against ovarian cancer cell cultures.
  Serum CA125 is commonly used as a tumor marker for ovarian cancer, and since it increases at a high rate in endometriosis, it has an aspect of being used as a diagnostic aid for endometriosis.
  There are many reports that the normal value of serum CA-125 is 35 U/mL or less.
  The test was performed during a non-menstruation period, as serum CA-125 levels are high during the menstrual period.
Time Frame: Baseline, and 5 months.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Cycle -1 | Cycle 5
Number analyzed (Participants) | 56 | 33
U/mL | 55.66 (70.57) | 47.52 (47.37)

8. Secondary Outcome: Change Over Time in Dysmenorrhea Score (Total of the Dysmenorrhea Severity Score and the Analgesic Use Score), Difference From Baseline
Description: The dysmenorrhea score is the sum of the dysmenorrhea severity score and the analgesic use score.
  The difference from baseline were calculated on an individual basis and these were totalled and means ± SD calculated.
  A dysmenorrhea severity score is defined as follows. None: Score 0, Rarely interfering with work (study and house work): Score 1, Interfering with work (study and house work) requiring lying down to rest: Score 2, Being confined to bed for 1 day, being unable to work (study and house work): Score 3.
  A score for the use of analgesics is defined as follows. None: Score 0, An analgesic was used for a day during the last (or current) menstruation period: Score 1, An analgesic was used for 2 days during the last (or current) menstruation period: Score 2, An analgesic was used for 3 days during the last (or current) menstruation period: Score 3
Time Frame: Baseline, 1 month, 2 months, 3 months, 4 months, and 5 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3 | Cycle 4 | Cycle 5
Number analyzed (Participants) | 57 | 52 | 50 | 45 | 42
score on a scale | -0.54 (1.45) | -0.90 (1.61) | -1.02 (1.30) | -0.96 (1.28) | -1.00 (1.47)
Statistical Analysis 1: Comparison: Cycle 1; The score value and difference from the value before treatment were calculated at the same points using the summary statistics, and the Wilcoxon signed-rank test was performed; Test type: Superiority; p = 0.0020, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cycle 2; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cycle 3; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cycle 4; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cycle 5; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change Over Time in Visual Analogue Scale (VAS) for Dysmenorrhea, Difference From Baseline
Description: A straight line with a total length of 10 cm was prepared. This straight line was defined as "no pain" at the left end and "Worst pain imaginable" at the right end.
  The cases marked the degree of pain on this straight line at each time point, and the length (cm) from the left end of the line (0) was measured.
  The minimum value of VAS is 0 cm (no pain) and the maximum value is 10 cm (Worst pain imaginable).
  The units on a scale is "cm". The difference from baseline were calculated on an individual basis and these were totalled and means ± SD calculated.
Time Frame: Baseline, 1 month, 2 months, 3 months, 4 months, and 5 months.
Population: One patient had a pain score at Cycle 1 but did not have a pain score at baseline and the absolute change could not be calculated in this instance
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3 | Cycle 4 | Cycle 5
Number analyzed (Participants) | 52 | 41 | 43 | 39 | 35
cm | -0.93 (2.24) | -1.61 (2.11) | -1.98 (2.38) | -1.94 (2.82) | -1.52 (2.18)
Statistical Analysis 1: Comparison: Cycle 1; The difference from the value before treatment and change rate were calculated using the summary statistics at each observation point and last observation, and the Wilcoxon signed-rank test was performed for the difference and change rate; Test type: Superiority; p = 0.0024, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cycle 2; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cycle 3; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cycle 4; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cycle 5; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change Over Time in Visual Analogue Scale (VAS) for Dysmenorrhea, Change Rate From Baseline (%)
Description: A straight line with a total length of 10 cm was prepared. This straight line was defined as "no pain" at the left end and "Worst pain imaginable" at the right end.
  The cases marked the degree of pain on this straight line at each time point, and the length (cm) from the left end of the line (0) was measured.
  The minimum value of VAS is 0 cm (no pain) and the maximum value is 10 cm (Worst pain imaginable).
  The change rate from baseline were calculated on an individual basis and these were totalled and means ± SD calculated.
Time Frame: Baseline, 1 month, 2 months, 3 months, 4 months, and 5 months.
Population: A number of patients at each timepoint had pain scores of "zero" or discontinued treatment and a % change could not be calculated in these instances
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cycle 1 | Cycle 2 | Cycle 3 | Cycle 4 | Cycle 5
Number analyzed (Participants) | 47 | 37 | 39 | 34 | 31
percent change | -9.23 (95) | -33.97 (65.48) | -38.01 (80.00) | -41.24 (76.62) | -35.75 (79.68)
Statistical Analysis 1: Comparison: Cycle 1; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0037, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Cycle 2; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Cycle 3; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Cycle 4; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Cycle 5; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0003, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Change in Serum CA125, Difference From Baseline
Description: The difference from baseline were calculated on an individual basis and these were totalled and means ± SD calculated.
  For the mean value of the difference shown here, the mean value of the difference of the cases that could be measured at each time point is calculated.
  In other words, of the 56 cases with baseline serum CA125, cycle 5 can only calculate the difference in 32 cases with serum CA125 at this point.
  The mean difference between cycle 5 and baseline in these 32 cases is shown here.
  The remaining 24 cases in Baseline are excluded from this calculation because they do not have serum CA125 measurements in Cycle 5.
  For this reason, these values cannot be calculated directly from the serum CA125 mean value at each time point shown in the result measurement 7.
Time Frame: Baseline, and 5 months.
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Cycle 5
Number analyzed (Participants) | 32
U/mL | -6.47 (97.38)
Statistical Analysis 1: Comparison: Cycle 5; Separately in the "efficacy analysis set" and "study completers," the values before treatment initiation and at last observation were compared, the value, difference from the value before treatment and change rate were calculated using the summary statistics, and the Wilcoxon signed-rank test was performed for the difference and change rate; Test type: Superiority; p = 0.8035, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Change in Serum CA125, Change Rate From Baseline (%)
Description: The change rate from baseline were calculated on an individual basis and these were totalled and means ± SD calculated.
  For the mean value of the change rate shown here, the mean value of the change rate of the cases that could be measured at each time point is calculated.
  In other words, of the 56 cases with baseline serum CA125, cycle 5 can only calculate the change rate in 32 cases with serum CA125 at this point.
  The mean change rate between cycle 5 and baseline in these 32 cases is shown here.
  The remaining 24 cases in baseline are excluded from this calculation because they do not have serum CA125 measurements in Cycle 5.
  For this reason, these values cannot be calculated directly from the serum CA125 mean value at each time point shown in the result measurement 7.
Time Frame: Baseline, and 5 months.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cycle 5
Number analyzed (Participants) | 32
percent change | 38 (183.02)
Statistical Analysis 1: Comparison: Cycle 5; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.8185, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: AE information during the survey was collected during a period from the start of Duphaston treatment to the end of the observation period or discontinuation. Approximately 5 months in the study completers.(From date of dosage start, up to 5 months)
Description: An adverse event (AE) is any unfavorable and unintended sign (including an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered causally related to the drug. If an AE was noted, a follow-up investigation was performed until it resolved whenever possible. AE information during the survey was collected during a period from the start of Duphaston treatment to the end of the observation period or discontinuation.
Groups:
- Dydrogesterone: Dydrogesterone 20 mg (4 tablets) per day should be orally administered in 2 divided doses (in the morning and evening). It should be administered for 21 days; dosage starts on the 5th day of each menstrual cycle until 25th day. The administration period will be from the start of Duphaston treatment (cycle 1) to cycle 4.
  Of 60 subjects whose case report forms were collected, 59 subjects were included in the "safety analysis set," after excluding one subject (reason: one subject, no data entered).
Arm/Group | Dydrogesterone
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 1/59
Other Adverse Events (participants affected / at risk) | 7/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dydrogesterone (N=59)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dydrogesterone (N=59)
Constipation (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Menstruation irregular (Reproductive system and breast disorders) | 1
Metrorrhagia (Reproductive system and breast disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT02921763/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/63/NCT02921763/SAP_001.pdf